CLINICAL TRIAL: NCT00781417
Title: Prevention of Secondary Hyperparathyroidism With Vitamin D in Stage II/III Chronic Kidney Disease
Acronym: POSH-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlanta VA Medical Center (U.S. Federal Agency)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Vin Tangpricha, Associate Professor, Atlanta VA Medical Center
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: Atlanta VAMC
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Kidney Disease
Keywords: vitamin D; Chronic Kidney Disease; parathyroid hormone; Chronic kidney disease Stage II and III
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Cholecalciferol 50,000 IU once a week for 12 weeks then every other week for 40 weeks
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — 50,000 IU once a week for 12 weeks then every other week for 40 weeks
  Other Names: cholecalciferol; vitamin D3
  Arms: 1
Other: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate whether earlier intervention with vitamin D in stage II/III chronic kidney disease will prevent or delay secondary hyperparathyroidism. Subjects will receive vitamin D or placebo at study entry and will be followed for a period of one year. The hypothesis is that subjects given vitamin D will have lower PTH and higher 25(OH)D after 1 year compared to placebo. Additionally, there will be less subjects who progress into secondary hyperparathyroidism in the vitamin D treated group compared to the placebo treated group.

DETAILED DESCRIPTION:
Vitamin D is important to maintain normal calcium homeostasis and optimal bone health (1, 2). The synthesis of vitamin D and its metabolism to 1,25(OH)2D is regulated by parathyroid hormone (PTH), serum calcium, and phosphorus levels. In response to low serum calcium level, serum PTH activates alpha-1-hydroxylase for increased 1,25(OH)2D production in the kidney and also enhances tubular reabsorption of calcium (3). The higher levels of 1, 25(OH)2D results in increased intestinal calcium absorption (4). Increased serum phosphorus levels which occurs in the early stages of chronic kidney disease (CKD) results in inhibition of the 1-alpha-hydroxylase, which results in decreased 1, 25(OH)2 D production, decreased intestinal calcium absorption leading to secondary hyperparathyroidism with increased PTH levels. Circulating 1,25(OH)2D levels begin to fall when the glomerular filtration rate is less than 40 mL/min occasionally even less than 80 mL/min (11) and almost always significantly reduced in subjects with end-stage renal failure (12). Furthermore, in CKD, decreased renal mass also results in decreased expression of 1-alpha-hydroxlase and less production of 1,25(OH)2D which also exacerbates secondary hyperparathyroidism (5-7).

Therefore, in CKD there are three processes that lead to secondary hyperparathyroidism. 1) decreased renal mass leading to decreased production of 1,25(OH)2D leading to a compensatory rise in PTH to further enhance production of 1,25(OH)2D 2) inhibition of the renal 1-alpha-hydroxylase by accumulating phosphorus levels leading to decreased 1,25(OH)2D which also leads to secondary hyperparathyroidism. 3) increased phosphorus leads to lower ionized calcium leading to increased parathyroid hormone secretion.

Untreated secondary hyperparathyroidism can lead to renal osteodystrophy (9) and increased mortality due to cardiovascular disease (10). Prolonged secondary hyperparathyroidism can lead to bone resorption and eventually autonomous parathyroid hormone secretion termed tertiary hyperparathyroidism.

Vitamin D status is one of the major factors that may prevent progression of secondary hyperparathyroidism in patients with CKD. Insufficient levels of 25-hydroxyvitamin D further exacerbate secondary hyperparathyroidism by not providing adequate substrate for the renal 1-alpha-hydroxylase for conversion to the active form of vitamin D, 1,25(OH)2D. A recent cross-sectional study on patients with moderate to severe CKD not yet on dialysis therapy from 12 geographically diverse regions of the United States has shown that only 29% and 17% of them had sufficient level, respectively (13). Vitamin D status is easily corrected. In our previous study we concluded that weekly cholecalciferol supplementation was an effective treatment to correct vitamin D status in patients with CKD stages III and IV (14). However, PTH levels did not return to normal. Therefore, it is likely that earlier intervention with vitamin D is necessary to prevent rather than to treat secondary hyperparathyroidism. This is the major question that is being evaluated in this study. Can intervening with vitamin D at an earlier stage of chronic kidney disease result in decreased incidence of secondary hyperparathyroidism?

2.0 Objectives

2.1 Overall Objective

The primary objective of this study is to assess that if improving and maintaining an optimal 25(OH) D level ( by National Kidney Foundation should be greater than 30ng/ml) (15) in people with stage II/III Chronic Kidney disease would delay the progression of secondary hyperparathyroidism and translate into improved markers of bone turnover

2.2 Specific Aims

Primary: 1) To determine in a double blind, randomized study whether supplementation with 50,000 IU of cholecalciferol (vitamin D3) given weekly for 12 weeks followed by maintenance cholecalciferol 50,000 IU every other week would improve and maintain vitamin D status in CKD patients stage 2/3 compared to placebo at 12 months.

2) To determine whether early intervention with vitamin D therapy further decreases PTH levels after 12 weeks of therapy and 12 months of therapy.

Secondary: 1) To determine whether early treatment with vitamin D results in improving levels of bone turnover markers- tartrate-resistant acid phosphatase isoform 5b(TRAP5b), procollagen Type 1 N-Terminal propeptide (PINP), serum C-Telopeptide and Alkaline phosphatase.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects must be patients with CKD stage II/III (estimated glomerular filtration rate, 30-90 ml/min/1.73m body surface area), 25-hydroxyvitamin D (25(OH) D) level >10 ng/ml documented in the medical record for the past 6 months.

Estimated Glomerular Filtration Rate will be calculated by using the original Modification of Diet in Renal Disease Study equation (online at http://www.nkdep.nih.gov)(16)

* Study subjects must agree to participate in the study and provide written informed consent
* Histology: not applicable
* Sites: Atlanta VA Medical Center
* Stage of Disease: CKD stage II/III, who has 25-hydroxyvitamin D (25(OH)D) level >10 ng/ml, but less than 30 ng/ml
* Age: Study subjects must be >18 but <85 years old
* Performance Status: Study subjects will be patients with CKD stage II/III (estimated glomerular filtration rate, 30-90 ml/min/1.73m body surface area), 25-hydroxyvitamin D (25(OH)D) level >10 ng/ml, but less than 30 ng/ml
* Informed consent requirements: All study subjects must agree to participate in the study and provide written informed consent, which will be written in English.

Exclusion Criteria:

* Age < 18years or >85 years old
* Prior other diseases: History of liver failure (AST or ALT >3 ULN), history of intestinal malabsorption or chronic diarrhea, corrected serum calcium >10.5 mg/dl, calcium x phosphorus product >70,treatment with more than 1000 IU of vitamin D per day; or current treatment with a vitamin D analogue or calcimimitec, taking antiepileptic medication, or other medications that could alter vitamin D metabolism(eg, phenytoin, phenobarbital, rifampin(17)
* Infection: not applicable

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-10; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
25(OH)D | 52 weeks
Parathyroid Hormone | 52 weeks
24 hour urine calcium | 52 weeks

SECONDARY OUTCOMES:
Markers of bone turnover | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vin Tangpricha, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Atlanta VAMC, Atlanta, Georgia, United States